CLINICAL TRIAL: NCT06722287
Title: Mobile Application for Early Detection and Intervention to Reduce Psychological Distress in Informal Family Caregivers of Community-dwelling Adults with Chronic Disorders in Thailand
Brief Title: Mobile Intervention for Mental Health of Family Caregivers in Thailand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Hongtu Chen, Research Scientist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023P001212; 5R21MH131043-02 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Depressive Symptoms, Generalized Anxiety, or Psychological Stress
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: 20 family caregivers will be asked to utilize each of the five CAMMA intervention components over a five-week period (i.e., about one component per week). At the initial home visit, research staff will set up network configuration (e.g., WiFi) and demonstrate step-by-step guidelines for using the features on the smartphone. The caregiver will then be asked to perform these tasks, to ensure that they have understood the instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAMMA Intervention (Experimental): Mobile application intervention that provides family caregivers with self-care tools, care management tools, and online support group
  Interventions: Behavioral: Caregiver Mental Health Mobile Application Intervention

INTERVENTIONS:
Behavioral: Caregiver Mental Health Mobile Application Intervention — The mobile application includes self-care tools, caregiving management tools, and online support groups

SUMMARY:
The goal of the R21 project is to develop a culturally informed Caregiver Mental Health Mobile Application program that will promote early detection of mental health problems and deliver an evidence-based self-care intervention for family caregivers providing care to adults with chronic disease in Thailand.

DETAILED DESCRIPTION:
The goal of the 2-year R21 project is to develop a culturally informed Caregiver Mental Health Mobile Application (hereafter referred to as CAMMA) program that will deliver an evidence-based intervention to reduce mental health problems in family caregivers of adults with chronic disorders in Thailand. Specific aims include: 1) Conducting qualitative research on family caregivers of persons with chronic disorders, focusing on their experience with mental health problems, caregiving practice, coping mechanisms, and socio-technological barriers to technology acceptance and use; 2) Develop a mobile application for the delivery of the CAMMA intervention; and 3) Conduct a formative evaluation of the CAMMA Intervention Components to ensure acceptability and usability of individual intervention components.

ELIGIBILITY:
Inclusion Criteria:

* adult (age 18 +) family caregiver (CG)
* has a minimum of 4 months of experience as a caregiver and provides at least 4 hours a day of care to the care recipient (CR);
* screen positive on depressive symptoms (score above 5 on PHQ-9), or generalized anxiety (score above 3 on GAD-2), or stress measured with Perceive Stress Scale (score above 6 on PPS-4)
* Access to a mobile device with internet access

Exclusion Criteria:

* Caregiver who refuses to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Usability | 5 weeks of intervention
  Measured by the System Usability Scale
Acceptability | 5 week of intervention
  Measured by the User Experience Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Public Health, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We need to decide on specific procedures and types of researchers for sharing the IPD.